CLINICAL TRIAL: NCT07282964
Title: Mindful Moms, Mindful Meals (MMMM): A Patient-Oriented Randomized Controlled Trial Testing the Effects of a Mindful Eating Intervention on Infant Feeding Practices
Brief Title: Mindful Moms, Mindful Meals (MMMM) Study
Acronym: MMMM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Brunswick (Other)
Responsible Party: Principal Investigator, Maryam Kebbe, Associate Professor, University of New Brunswick
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB 2025-126
Record Dates: First submitted 2025-09-12; First posted 2025-12-15 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-12

CONDITIONS: Nutrition in Early Infancy; Nutrition Habits; Postpartum Nutrition; Mindful Eating Intervention
Keywords: Infant; Feeding Behavior; Postpartum Period; Diet; Mindful Eating; Nutrition
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Intervention Model Description: Parallel Waitlist-Control Randomized Controlled Trial
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants in this group will take part in an 8-week, tailored Mindfulness-Based Eating Awareness Training Postpartum (MB-EAT-P) program. Weekly sessions will include mindfulness meditations, training in hunger and satiety awareness, responsive feeding education, light-intensity physical activity, and food tasting experiences. In addition to the group sessions, participants will be encouraged to engage in at-home practices, including mindfulness meditations, mindful eating, responsive feeding techniques, and journaling their experiences to support reflection and integration of the training into daily life.
  Interventions: Behavioral: Mindfulness-Based Eating Awareness Training Postpartum
- Control (Active Comparator): Participants in the control group will receive access to the Mindfulness-Based Eating Awareness Training Postpartum (MB-EAT-P) program following the initial 8-week period. This self-guided version of the program will be delivered through the MMMM website and will include recorded sessions, meditation scripts, worksheets, and all core components of the intervention. These components encompass mindfulness meditations, hunger and satiety awareness training, responsive feeding education, light-intensity physical activity guidelines, and food tasting guidance.
  Interventions: Behavioral: Waitlist Mindfulness-Based Eating Awareness Training Postpartum

INTERVENTIONS:
Behavioral: Mindfulness-Based Eating Awareness Training Postpartum — Mindfulness-Based Eating Awareness Training Postpartum (MB-EAT-P) is an 8-week, patient-oriented intervention co-developed with a Parent Advisory Committee. Designed for postpartum individuals, it integrates mindfulness practices, responsive feeding education, and experiential learning. Weekly sessions include guided meditations, mindful eating exercises, infant feeding strategies, and reflective journaling. Activities cover hunger/satiety cues, emotional balance, cultural feeding practices, and light physical activity. MB-EAT-P stands out for its postpartum-specific design, parent-led development, and holistic approach to maternal-infant well-being.
  The intervention group receives the full program following the baseline visit, in an in-person group setting.
  Arms: Intervention
Behavioral: Waitlist Mindfulness-Based Eating Awareness Training Postpartum — Mindfulness-Based Eating Awareness Training Postpartum (MB-EAT-P) is an 8-week, patient-oriented intervention co-developed with a Parent Advisory Committee. Designed for postpartum individuals, it integrates mindfulness practices, responsive feeding education, and experiential learning. Weekly sessions include guided meditations, mindful eating exercises, infant feeding strategies, and reflective journaling. Activities cover hunger/satiety cues, emotional balance, cultural feeding practices, and light physical activity. The control group will not receive any components of the intervention until after the final clinical visit. MB-EAT-P stands out for its postpartum-specific design, parent-led development, and holistic approach to maternal-infant well-being.
  The control group will then receive the full program post-study via the MMMM website in a self-guided format with recorded sessions, scripts, and worksheets.
  Arms: Control

SUMMARY:
The goal of this clinical trial is to learn whether a Mindfulness-Based Eating Awareness Training Postpartum (MB-EAT-P) program can improve infant feeding practices and maternal eating behaviors. Researchers will compare participants who receive the MB-EAT-P program immediately to those who receive it after an 8-week waitlist period. Participants in the intervention group will attend weekly 2-hour MB-EAT-P sessions for 8 weeks and practice mindfulness and mindful eating at home. Participants in both groups will participate in a recorded mealtime observations with their infant and complete surveys and dietary recalls at baseline, midpoint, and post-intervention. This study is patient-oriented and co-developed with a Parent Advisory Committee to ensure relevance to postpartum individuals.

DETAILED DESCRIPTION:
Background. Postpartum life may lead to suboptimal nutrition behaviors/habits. Mothers have reported an unbalanced diet postpartum, defined as insufficient intake of key food groups i.e., fruits, veggies, grain foods, dairy and meat, which is directly linked to obesity, diabetes, and cancer. Maternal eating behaviours also contribute to child feeding practices, which in turn shape their lifelong eating patterns. Mindful eating can help struggling mothers to re-balance their nutrition by increasing awareness of choices, reducing stress, and fostering a greater connection to bodily cues, such as hunger and fullness cues. Previous literature on mindful eating has focused on the pregnant population and found that mindfulness-based interventions are feasible and acceptable, can reduce stress and overeating during pregnancy, and may support healthier postpartum weight outcomes through intuitive eating practices. The effects of postpartum mindful eating interventions on mothers' diet and feeding of infants remain unknown.

Objectives. The Mindful Moms, Mindful Meals (MMMM) study aims to evaluate the effects of a Mindfulness-Based Eating Awareness Training Postpartum (MB-EAT-P) intervention on infant feeding practices and maternal eating behaviors.

Research Questions.

* Does MB-EAT-P improve mothers' recognition of infant hunger and satiety cues?
* Does MB-EAT-P enhance maternal mindful eating?
* Does MB-EAT-P improve dietary quality of mother and infant?
* Does MB-EAT-P improve behaviour change constructs (e.g., knowledge, confidence, self-efficacy?)
* Does MB-EAT-P improve sleep quality, weight control, and anxiety symptoms?
* Does MB-EAT-P promote sustainable mindful eating and responsive feeding behaviours 3-months post-intervention?

Methodological Approach. This parallel, waitlist-control randomized controlled trial will adapt an 8-week mindful eating intervention for postpartum participants. Approximately 72 participants, aged 19-45 years, with infants aged 6-12 months who have started solid foods, will be recruited from social media, community outreach, and local health clinics in Fredericton, NB. Exclusion criteria include active eating disorders, substance use disorders, unmanaged medical/mental health conditions such as diagnosed postpartum depression or anxiety, cognitive impairments, recent trauma or untreated post-traumatic stress disorder, participation in a similar program within 12 months, strict dietary regimens, recent major surgery that affects nutritional intake, preterm infants, or no English proficiency.

Mothers will be randomized to either the intervention group or a control group using REDCap®. The intervention group will begin the MB-EAT-P program immediately upon enrollment, participating in 2-hour weekly group sessions over eight weeks, guided by MB-EAT certified instructor, with supplemental at-home mindfulness practices. Sessions will cover topics such as transitioning from breastfeeding and formula-feeding to solid foods, hunger and satiety awareness, recognition and management of emotional and mindless eating, and mindful eating strategies tailored for the postpartum period, including infancy. Meanwhile, the control group will be waitlisted for eight weeks. After the waitlist period, the control group will receive the intervention materials via the MMMM website, including recordings of guided mindful eating meditations, session worksheets, and responsive feeding infographics.

Phenotypic assessments will occur at the University of New Brunswick by telephone and/or online. Data will be collected at baseline, 4 weeks (midpoint), 8 weeks (post-intervention) and 3-months post-intervention. Infant feeding practices will be observed, using the validated Responsiveness to Child Feeding Cues Scale, during a recorded individual mealtime session in the PEADS Lab Metabolic Kitchen. The Mindful Eating Scale (MES) and Mindful Eating Behavior Scale (MEBS) will measure maternal mindful eating. Other questionnaires will measure maternal and infant feeding, weight control strategies, sleep, and mental health. Dietary quality of mothers and infants will be measured using the Healthy Eating Food Index and the WHO Infant and Young Child Feeding Indicators, respectively, derived from a 24-hour dietary recall.

Infant feeding practices, maternal eating behaviours, and dietary quality are among the top priorities for mothers. Our outcomes draw from this literature, as well as the priorities identified by moms in our Parent Advisory Committee (PAC). Specifically, the investigators established a PAC consisting of five diverse postpartum mothers from across Canada following the Canadian Institutes for Health Research recommendations for patient engagement. PAC mothers have collaborated (level 4 of 5 of the IAP2) with the research team by contributing to the development of MB-EAT-P session materials as well as informed session timings, postpartum specific programming, MMMM website and child-minding volunteer program.

Statistical Analysis. A repeated measures analysis of covariance (ANCOVA) will be conducted to evaluate the interaction between time (three measurements) and group (intervention vs. control). Based on a repeated measures within-between group interaction (ie. whether the pattern of change over time differs between groups), and assuming a small-to-medium effect size (f = 0.2), α = 0.05, and 95% power, 66 participants (28 per group) are required; to account for an anticipated ~10% drop-out rate, 72 participants (36 per group) will be recruited. A comprehensive analysis of 32 studies reported pooled effect sizes ranging approximately from f = 0.11 to f = 0.35, indicating small to moderate improvements in mindless eating behaviors such as controlled eating, fullness awareness, and impulsive food choices. The effects on stress-related eating behaviors, including emotional and binge eating, were generally smaller and less consistent across studies. However, an effect size of f = 0.32 for fullness awareness and f = 0.25 for long-term improvements in hunger eating were reported in adults, reflecting a medium-sized effect in the context of mindful eating interventions, suggesting an f = 0.20 for MMMM is appropriate yet conservative for an infant population.

Expected Outcomes. This study will generate evidence on how mindful eating interventions, like MB-EAT-P, may enhance maternal and infant feeding practices. Our findings may inform the development of public health programs to promote lifelong mindful eating and feeding habits.

ELIGIBILITY:
Inclusion Criteria:

* Age between 19 and 45 years.
* Have started or plan to start solid foods for their baby by the time of enrollment
* Have an infant aged 6 to 12 months
* Willing to participate in a recorded mealtime observation for the study
* Willing to complete an 8-week MB-EAT-P intervention, including homework assignments
* Have an infant born at or after 37 weeks of gestation.

Exclusion Criteria:

General

* Planning to move in the next two months
* Medically diagnosed with an active eating disorder (e.g., Anorexia, Bulimia, Binge Eating Disorder)
* Diagnosed with an unmanaged chronic medical condition affecting diet (e.g., uncontrolled diabetes, celiac disease, severe GI disorders, kidney disease, sleep apnea, PCOS)
* Diagnosed with unmanaged postpartum depression or anxiety
* Diagnosed with iron-deficiency anemia with extreme fatigue or weakness
* Substance use disorder (e.g., alcohol or drug addiction)
* Cognitive impairments affecting memory, attention, or comprehension (e.g., dementia, brain injury)
* Following a strict formal diet or weight loss program
* Enrolled in a weight loss or mindfulness-based program in the past 12 months
* Recovering from major surgery or experiencing an acute medical crisis (e.g., bariatric surgery)
* Experiencing recent trauma or untreated PTSD

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Infant Responsive Feeding | Baseline, at 4 weeks, at 8 weeks after enrollment and 3 months post-intervention
  Responsive Feeding is defined as a caregiver's ability to recognize and appropriately respond to their infant's hunger and satiety cues in a timely, supportive, and developmentally appropriate manner. It includes offering food when the infant shows hunger, allowing self-regulation, and avoiding coercive feeding. Infant cues will be assessed using the Responsiveness to Child Feeding Cues Scale (RCFCS), an observational coding system rating hunger and satiety cues (early, active, late), engagement, affect, and physical disposition. Cue strength is rated 1-5, with late cues coded present (1), absent (0), or can't tell (6). Responsiveness reflects how accurately and promptly caregivers respond to these cues, rather than cue strength alone. Composite measures include infant receptiveness (balance of hunger vs. fullness cues) and feeding engagement (percentage of time engaged with feeding). Trained coders will code video-recorded meals using the standardized RCFCS manual.
Maternal Mindful Eating | Baseline, at 4 weeks, at 8 weeks after enrollment and 3 months post-intervention
  Mindful Eating is defined as non-judgmental awareness of physical and emotional sensations during eating, including hunger, satiety, taste, and emotional triggers. In this study, maternal mindful eating will be assessed using two validated tools: the Mindful Eating Questionnaire (MEQ) and the Mindful Eating Behavior Scale (MEBS). The MEQ evaluates dimensions such as awareness, disinhibition, and emotional eating, with scores ranging from 1 to 4, where higher scores reflect more mindful eating. The MEBS measures behavioral engagement in mindful eating practices, with scores from 1 to 5, with higher scores indicating greater mindful eating behavior. Together, the MEQ and MEBS provide a multidimensional understanding of how postpartum individuals engage with food and feeding in a mindful, intentional way, capturing both attitudinal and behavioral aspects of mindful eating.

SECONDARY OUTCOMES:
Dietary Quality | Baseline, at 4 weeks, and at 8 weeks after enrollment.
  Dietary quality is defined as the overall nutritional adequacy and alignment of food intake with dietary guidelines. Maternal dietary quality will be assessed using the Healthy Eating Food Index (HEFI) based on ASA24 dietary recalls, which evaluates intake across food groups and nutrients. HEFI scores range from 0 to 80, with higher scores reflecting better alignment with recommendations. Infant dietary quality will be assessed using the WHO Infant and Young Child Feeding (IYCF) Indicators, which capture dietary diversity (0-7 food groups), meal frequency, and breastfeeding status. Together, the HEFI and IYCF provide a comprehensive assessment of maternal and infant nutritional behaviors and adherence to recommended feeding standards.
Behaviour Change Constructs | Baseline, at 4 weeks, and at 8 weeks after enrollment.
  The investigators will examine whether MB-EAT-P improves behaviour change constructs (e.g., knowledge, confidence, self-efficacy) assessed using the Maternal Self-Efficacy Questionnaire for Solid Feeding (MSEQ-SF) and the InFANT Program Questionnaire. The MSEQ-SF captures maternal confidence and self-efficacy across three domains: (1) responsive feeding (ability to recognize hunger/satiety cues; range 0-20), (2) capability to feed (providing healthy food and encouraging intake; range 5-25), and (3) food-related decisions (confidence in making appropriate feeding choices; range 0-8). The InFANT Program Questionnaire assesses nutrition knowledge (12 items scored on a 4-point agreement scale, dichotomized into correct/incorrect) and parental confidence in promoting healthy eating, limiting unhealthy foods, and providing healthy settings (scored on a 5-point confidence scale).
Sleep Quality | Baseline, at 4 weeks, and at 8 weeks after enrollment.
  The investigators will examine whether MB-EAT-P improves sleep quality in mothers. Sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI). The PSQI total score ranges from 0 to 21, with higher scores indicating poorer sleep quality.
Weight Control Strategies | Baseline, at 4 weeks, and at 8 weeks after enrollment.
  The investigators will examine whether MB-EAT-P improves weight control strategies. Weight control strategies will be assessed using the Weight Control Strategies Scale (WCSS). The WCSS includes subscales for dietary choices, self-monitoring, and physical activity, with scores ranging from 0 to 4 per item; higher scores indicate more frequent use of weight control strategies.
Mental Health | Baseline, at 4 weeks, and at 8 weeks after enrollment.
  The investigators will examine whether MB-EAT-P improves mental health symptoms such as postpartum anxiety. Mental health will be assessed using the Symptom Checklist-90 (SCL-90). The SCL-90 contains 90 items scored from 0 to 4, producing subscale scores (e.g., Depression, Anxiety, Somatization) and a Global Severity Index (GSI); higher scores indicate greater psychological distress.
Sustainability of Mindful Eating | 3 months post-intervention
  Self-Regulation of Eating Behaviour Questionnaire (SREBQ) will be administered 3 months post intervention to assess sustainability of Mindful Eating behaviours. SREBQ is scored on a scale of 1-5 for five questions. The score ranges between 25-5 with higher score indicating better self-regulation of Mindful Eating Behaviour.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Maryam Kebbe, PhD, CLC, Principal Investigator — University of New Brunswick
Locations (1):
- University of New Brunswick, Fredericton, New Brunswick, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kao TA, Ling J, Alanazi M, Atwa A, Liu S. Effects of mindfulness-based interventions on obesogenic eating behaviors: A systematic review and meta-analysis. Obes Rev. 2025 Mar;26(3):e13860. doi: 10.1111/obr.13860. Epub 2024 Nov 3. PMID 39489689
- [Background] Ayyala MS, Coughlin JW, Martin L, Henderson J, Ezekwe N, Clark JM, Appel LJ, Bennett WL. Perspectives of pregnant and postpartum women and obstetric providers to promote healthy lifestyle in pregnancy and after delivery: a qualitative in-depth interview study. BMC Womens Health. 2020 Mar 4;20(1):44. doi: 10.1186/s12905-020-0896-x. PMID 32131832
- [Background] Madray C, Richardson J, Hornsby P, Grello C, Drake E, Kellams A. Exploring the Unmet Needs of Postpartum Mothers: A Qualitative Study. J Perinat Educ. 2022 Apr 1;31(2):71-81. doi: 10.1891/JPE-2021-00009. PMID 35386495
- [Background] Brassard D, Elvidge Munene LA, St-Pierre S, Guenther PM, Kirkpatrick SI, Slater J, Lemieux S, Jessri M, Haines J, Prowse R, Olstad DL, Garriguet D, Vena J, Vatanpatast H, L'Abbe MR, Lamarche B. Development of the Healthy Eating Food Index (HEFI)-2019 measuring adherence to Canada's Food Guide 2019 recommendations on healthy food choices. Appl Physiol Nutr Metab. 2022 May;47(5):595-610. doi: 10.1139/apnm-2021-0415. Epub 2022 Jan 14. PMID 35030038
- [Background] Manafo E, Petermann L, Vandall-Walker V, Mason-Lai P. Patient and public engagement in priority setting: A systematic rapid review of the literature. PLoS One. 2018 Mar 2;13(3):e0193579. doi: 10.1371/journal.pone.0193579. eCollection 2018. PMID 29499043
- [Background] Leahy K, Berlin KS, Banks GG, Bachman J. The Relationship Between Intuitive Eating and Postpartum Weight Loss. Matern Child Health J. 2017 Aug;21(8):1591-1597. doi: 10.1007/s10995-017-2281-4. PMID 28176035
- [Background] Ward K, Herekar A, Wang P, Lindsay KL. Feasibility and Acceptability of a Mindfulness-Based Smartphone App among Pregnant Women with Obesity. Int J Environ Res Public Health. 2023 Apr 6;20(7):5421. doi: 10.3390/ijerph20075421. PMID 37048035
- [Background] Vieten C, Laraia BA, Kristeller J, Adler N, Coleman-Phox K, Bush NR, Wahbeh H, Duncan LG, Epel E. The mindful moms training: development of a mindfulness-based intervention to reduce stress and overeating during pregnancy. BMC Pregnancy Childbirth. 2018 Jun 1;18(1):201. doi: 10.1186/s12884-018-1757-6. PMID 29859038
- [Background] Tylka TL, Eneli IU, Kroon Van Diest AM, Lumeng JC. Which adaptive maternal eating behaviors predict child feeding practices? An examination with mothers of 2- to 5-year-old children. Eat Behav. 2013 Jan;14(1):57-63. doi: 10.1016/j.eatbeh.2012.10.014. Epub 2012 Nov 10. PMID 23265403
- [Background] Roberts LT, Carbonneau N, Goodman LC, Musher-Eizenman DR. Retrospective reports of childhood feeding in mother-daughter dyads. Appetite. 2020 Jun 1;149:104613. doi: 10.1016/j.appet.2020.104613. Epub 2020 Jan 24. PMID 31987877
- [Background] Furman D, Campisi J, Verdin E, Carrera-Bastos P, Targ S, Franceschi C, Ferrucci L, Gilroy DW, Fasano A, Miller GW, Miller AH, Mantovani A, Weyand CM, Barzilai N, Goronzy JJ, Rando TA, Effros RB, Lucia A, Kleinstreuer N, Slavich GM. Chronic inflammation in the etiology of disease across the life span. Nat Med. 2019 Dec;25(12):1822-1832. doi: 10.1038/s41591-019-0675-0. Epub 2019 Dec 5. PMID 31806905
- [Background] Faria-Schutzer DB, Surita FG, Rodrigues L, Turato ER. Eating Behaviors in Postpartum: A Qualitative Study of Women with Obesity. Nutrients. 2018 Jul 10;10(7):885. doi: 10.3390/nu10070885. PMID 29996489
- See also: Infant and young child feeding. World Health Organization — https://www.who.int/data/nutrition/nlis/info/infant-and-young-child-feeding
- See also: Government of Canada CIHR. Patient engagement - CIHR — https://cihr-irsc.gc.ca/e/45851.html